CLINICAL TRIAL: NCT05114954
Title: A Prospective, Multicenter, Single-arm Objective Performance Criteria Evaluation of the Safety and Efficacy of a Pulsed Field Ablation System in Patients With Paroxysmal Atrial Fibrillation
Brief Title: Evaluation of the Safety and Efficacy of the CardioPulseTM PuLsed fiEld Ablation SystEm in Patients With Paroxysmal Atrial Fibrillation (PLEASE-AF Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Dinova EP Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFA001
Record Dates: First submitted 2021-10-21; First posted 2021-11-10 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment group (Experimental): Patients treated with PFA catheter.
  Interventions: Device: CardioPulsesTM pulsed field ablation system

INTERVENTIONS:
Device: CardioPulsesTM pulsed field ablation system — Using pulsed field ablation (PFA) catheter, steerable sheath and pulsed field generator to treat atria fibrillation.

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and efficacy of a pulsed field ablation system developed and manufactured by Hangzhou Dinova EP Technology Co., Ltd in the treatment of patients with paroxysmal atrial fibrillation

DETAILED DESCRIPTION:
This study is a premarket clinical trial of a pulsed field ablation catheter system, this study evaluates the safety and effectiveness of the pulsed field ablation catheter system developed and produced by Hangzhou Dinova EP Technology Co., Ltd. in the endovascular interventional treatment of patients with paroxysmal atrial fibrillation, and provided a clinical basis for the formal application of this product in China.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 75 years old;
2. Patients diagnosed with symptomatic paroxysmal atrial fibrillation:

   At least 1 ECG or rhythm monitoring documented AF episode within 12 months prior to enrollment.
3. Ineffective or intolerant of at least one antiarrhythmic drug;
4. Able to understand the purpose of the trial, participate in the trial voluntarily with informed consent form signed by the subject him/herself or his or her legal representative, and willing to complete follow-up visits as required under the protocol.

Exclusion Criteria:

1. AF secondary to electrolyte imbalance, thyroid disease, or reversible cause;
2. Persistent or long-standing persistent AF;
3. Previous surgery or catheter ablation for AF;
4. Participant known to require ablation outside the pulmonary vein or in cavotricuspid isthmus region (such as atrioventricular reentrant tachycardia, atrioventricular nodalreentry tachycardia, atrial tachycardia, atrial flutter, ventricular tachycardia and Wolff-Parkinson-White syndrome);
5. Previous valve repair, replacement or artificial valve implantation; previous atrial septal defect closure, patent foramen ovale closure cardiac intervention or surgery;
6. Previous left atrial appendage closure;
7. Any myocardial infarction (MI), coronary artery bypass grafting (CABG) procedure or percutaneous coronary intervention (PCI) during the 6-month interval preceding the consent date;
8. Any carotid artery stent implantation or endarterectomy within the previous 6 months;
9. Left atrial diameter≥50 mm (anteroposterior);
10. LVEF <40% on admission, or NYHA class III and IV;
11. Presence of implanted ICD, CRT, permanent pacemaker, or any type of implantable device
12. Documented active thrombus in the left atrium or atrial appendage on imaging;
13. Rheumatic heart disease;
14. Uncontrollable high blood pressure;
15. Hypertrophic cardiomyopathy, myocardial thickening was significantly greater than or equal to 15mm;
16. Frequent premature ventricular beats;
17. Documented thromboembolic event (including TIA) within the past 6 months;
18. Presence of intramural thrombus, tumor or other abnormality that precludes vascular access or catheter manipulation;
19. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gas or severe breathing difficulties;
20. Anticoagulation contraindications, and history of blood clotting or bleeding abnormalities;
21. Patients with acute systemic infection;
22. Serum creatinine is more than twice the upper normal limit, or have a history of kidney dialysis;
23. Women who are pregnant and/or breast feeding or unable to use contraception during the trial;
24. Enrollment in another clinical trial evaluating other devices or drugs during the same period;
25. Life expectancy less than 12 months (such as patients with advanced cancer);
26. Abnormalities or diseases that the investigator considers to be excluded from the study's coverage.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
The effectiveness of the pulsed field ablation system in the treatment of paroxysmal atrial fibrillation is evaluated by the 12-month ablation success rate of atrial fibrillation. | 12 months after the ablation
  12-month ablation success rate of atrial fibrillation is defined by ECG data (including ECG and 24-hour dynamic electrocardiogram (Holter)) during the effective evaluation period (blanking period to the end of 12-month follow-up), without recording AF, AFL or AT (Arrhythmia monitoring device ≥ 30 seconds).

SECONDARY OUTCOMES:
Acute isolation success rate | 20 minutes after the ablation
  Acute isolation success refers to maintaining electrical isolation of the pulmonary vein 20 minutes after completion of all pulmonary vein ablation.
Ablation efficiency including total procedure time, catheter dwell time, pulse discharge time and total X-ray exposure time | immediately after the ablation
  Total procedure time (defined as the total time from initial femoral venipuncture to final catheter removal), catheter dwell time (time between the pulsed field ablation catheter entering the left atrium and its withdrawal from the left atrium), pulse discharge time (The total time of delivering pulse energy through the pulsed field ablation catheter, single ablation time ablation times), total X-ray exposure time (the total time of X-ray imaging of the catheter).
Incidence of device-related or operating-related major adverse events (MAE) 3 months after surgery | 3 months after the ablation
  Including death, myocardial infarction, stroke or transient ischemic attack (TIA), pulmonary vein stenosis, phrenic nerve palsy, systemic circulatory embolism, pericarditis*, cardiac tamponade/perforation, atrial esophageal fistula, and severe vascular access complications.
Incidence of severe adverse events | 12 months after the ablation
  Refers to an event that occurs during the clinical trial that results in mortality or serious deterioration in patient health, including a fatal illness or injury, a permanent defect in body structure or body function, or an event that requires medical or surgical intervention to avoid one or more permanent defects in body structure or body function.
Incidence of device-related adverse events | 12 months after the ablation
  Device-related adverse events refer to an adverse medical event related to the use of a device that occurs during the course of the clinical trial. However, a distinction should be made with respect to normal postoperative stress response, such as fever and chest and back discomfort, which, in the judgment of the investigator, need not be recorded as an adverse event. Recording of device-related adverse events will be applicable for conditions that are deemed by the investigator to be definitely related, possibly related, or of indeterminate relationship, to the test device.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of the Northern Theater of the Chinese People's Liberation Army, Shenyang, China

REFERENCES:
- [Derived] Wang Z, Tang M, Reddy VY, Chu H, Liu X, Xue Y, Wang J, Xu J, Liu S, Xu W, Zhang Z, Han B, Hong L, Yang B, Ding M, Liang M. Efficacy and safety of a novel hexaspline pulsed field ablation system in patients with paroxysmal atrial fibrillation: the PLEASE-AF study. Europace. 2024 Jul 2;26(7):euae174. doi: 10.1093/europace/euae174. PMID 38912887